CLINICAL TRIAL: NCT01887106
Title: Randomized, Double-blind, Placebo-controlled, Dose-ranging Study for the Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Oral Doses of GLPG1205 in Healthy Male Subjects
Brief Title: First-in-Human Single and Multiple Dose of GLPG1205
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1205-CL-101
Record Dates: First submitted 2013-06-22; First posted 2013-06-26 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — Suspensions; GLPG1205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GLPG1205 single dose (Experimental): Single oral dose of GLPG1205 suspension - ascending doses
  Interventions: Drug: GLPG1205 single ascending doses, oral suspension
- Placebo single dose (Placebo Comparator): Single oral dose of placebo suspension
  Interventions: Drug: Placebo single ascending doses, oral suspension
- GLPG1205 multiple doses (Experimental): Multiple oral doses of GLPG1205 suspension - ascending doses
  Interventions: Drug: GLPG1205, multiple ascending doses, oral suspension
- Placebo multiple doses (Placebo Comparator): Multiple oral doses of placebo suspension
  Interventions: Drug: Placebo, multiple ascending doses, oral suspension

INTERVENTIONS:
Drug: GLPG1205 single ascending doses, oral suspension — Single dose, oral suspension at 10 mg/mL or 50 mg/mL, starting dose of 10mg escalating up to 800mg
  Arms: GLPG1205 single dose
Drug: Placebo single ascending doses, oral suspension — Single dose, oral suspension matching placebo
  Arms: Placebo single dose
Drug: GLPG1205, multiple ascending doses, oral suspension — Multiple doses, daily for 14 days, oral suspension at 10 mg/mL or 50 mg/mL, anticipated doses: 100mg to 400mg
  Arms: GLPG1205 multiple doses
Drug: Placebo, multiple ascending doses, oral suspension — Multiple doses, daily for 14 days, oral suspension matching placebo
  Arms: Placebo multiple doses

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety and tolerability after single ascending oral doses of GLPG1205 given to healthy male subjects, compared to placebo. Also, the safety and tolerability of multiple ascending oral doses of GLPG1205 given to healthy male subjects daily for 14 days compared to placebo, will be evaluated.

Furthermore, during the course of the study after single and multiple oral dose administrations, the amount of GLPG1205 present in the blood and urine (pharmacokinetics) as well as the receptor occupancy by GLPG1205 in blood samples (pharmacodynamics) will be characterized compared to placebo.

Also, the potential of cytochrome P450 (CYP)3A4 induction after repeated dosing with GLPG1205 will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 18-50 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability after single dose | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1205 in comparison with placebo after a single oral dose in healthy subjects in terms of adverse events, physical examinations, vital signs, ECG and lab assessments
Safety and tolerability after multiple doses | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG1205 in comparison with placebo after multiple oral doses daily for 14 days in healthy subjects in terms of adverse events, physical examinations, vital signs, ECG and lab assessments

SECONDARY OUTCOMES:
The amount of GLPG1205 in plasma and urine over time after a single oral dose | Between Day 1 predose and 48 hours post dose
  To characterize the amount of GLPG1205 in plasma and urine over time - pharmacokinetics (PK) - after a single oral dose in healthy subjects
The amount of GLPG1205 in plasma and urine over time after multiple oral doses | Between Day 1 predose and Day 16 (48 hours after the last dose)
  To characterize the amount of GLPG1205 in plasma and urine over time - pharmacokinetics (PK) - after multiple oral doses in healthy subjects
Ratio of 6-b-hydroxycortisol/cortisol in urine | Twelve hours before dosing on Day 1 and Day 14
  To assess the potential of CYP3A4 induction after repeated dosing with GLPG1205 by means of the ratio of 6-b-hydroxycortisol/cortisol in urine
Receptor occupancy by GLPG1205 on blood cells after a single dose | Day 1 predose up to 24 hours post dose
  To characterize the pharmacodynamics (PD) of GLPG1205 by means of receptor occupancy by GLPG1205 on blood cells after a single oral dose in healthy subjects
Receptor occupancy by GLPG1205 on blood cells after multiple doses | Day 1 and Day 14, predose up to 24 hours post dose
  To characterize the pharmacodynamics (PD) of GLPG1205 by means of receptor occupancy by GLPG1205 on blood cells after multiple oral doses in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium